CLINICAL TRIAL: NCT02699931
Title: A Randomized, Investigator-blinded, 3-month, Parallel Group Clinical Study to Compare the Efficacy of Electric 3D Toothbrushes Versus Manual Toothbrushes in Patients With Fixed Orthodontic Appliances
Brief Title: Efficacy of Electric 3D Versus Manual Toothbrushes in Patients With Fixed Orthodontic Appliances
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Demetrios Halazonetis, Assoc. Prof., National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2THBRUSH01
Record Dates: First submitted 2016-03-01; First posted 2016-03-07 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Gingivitis; Dental Plaque
MeSH Terms: conditions — Gingivitis; Dental Plaque

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electric3D (Experimental): 3D electric toothbrush (Oral-B) with orthodontic head.
  Interventions: Device: Electric3D
- Manual (Active Comparator): Manual orthodontic toothbrush (Oral-B).
  Interventions: Device: Manual

INTERVENTIONS:
Device: Electric3D — Oral-B 3D with orthodontic head
  Arms: Electric3D
Device: Manual — Oral-B orthodontic
  Arms: Manual

SUMMARY:
This study evaluates if electric toothbrushes with a 3D action (rotation / oscillation and pulsation) are more effective than manual toothbrushes in removing plaque and reducing gingival inflammation in patients under orthodontic treatment with fixed appliances.

DETAILED DESCRIPTION:
This trial is designed as a randomized, controlled, investigator blinded superiority trial, with two parallel groups and a 1:1 allocation ratio. Equal number of males and females will be allocated to each group.

One group of orthodontic patients will receive an electric toothbrush with orthodontic head and the other group will receive a manual orthodontic brush. Tooth brushing instructions will be provided. Measurements of two plaque indices and two gingival indices will be taken at baseline and at 3 monthly intervals.

ELIGIBILITY:
Inclusion Criteria:

- Age between 12 and 16 years. Good general health according to a recent full medical history. Fixed labial orthodontic appliances on all teeth from central incisor to first molar (bands on first molars, metallic brackets-conventional, not self ligating-on other teeth), in both the maxillary and the mandibular arch, placed at least two months before the patient is accepted into the study and no more than two years.

Non-extraction orthodontic treatment. Plaque-induced gingivitis: patients will be included if they have gingival bleeding on at least 30% of the sites examined using the criteria for bleeding of the Modified Simplified Gingival Index.

Exclusion Criteria:

- Active caries. Periodontitis. Tooth agenesis (excluding third molars). Syndromes and craniofacial deformities. Current use of electric toothbrush. More than two cervical and/or proximal fillings. Dental prostheses or dental implants. Smoking or use of other tobacco products. Antibiotics during the last 2 months. Medication that may result in gingival enlargement (e.g. anticonvulsants, immunosuppressants, calcium channel blockers).

Disabilities that might affect toothbrushing skills (manual dexterity, mental disabilities).

Peri-oral or intra-oral piercing. Cardiac or other medical condition that requires antibiotic prophylaxis for dental treatment.

Participation in other trials.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Modified Silness and Löe plaque index | Baseline and monthly for 3 months
Modified Full mouth plaque score | Baseline and monthly for 3 months
Modified Gingival index | Baseline and monthly for 3 months
Modified Simplified Gingival index | Baseline and monthly for 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Demetrios J Halazonetis, Principal Investigator — National and Kapodistrian University of Athens
Locations (1):
- Department of Orthodontics, School of Dentistry, Athens, Greece

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Mylonopoulou IM, Pepelassi E, Madianos P, Halazonetis DJ. A randomized, 3-month, parallel-group clinical trial to compare the efficacy of electric 3-dimensional toothbrushes vs manual toothbrushes in maintaining oral health in patients with fixed orthodontic appliances. Am J Orthod Dentofacial Orthop. 2021 Nov;160(5):648-658. doi: 10.1016/j.ajodo.2021.02.016. PMID 34752255